CLINICAL TRIAL: NCT00826072
Title: Association Study of Inflammatory Genetic Polymorphism and Acute Lung Injury After Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Inflammatory Genetic Polymorphism and Acute Lung Injury After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Jia-feng Wang, M.D., Changhai Hospital
Other Study IDs: PCSP-inflammation
Record Dates: First submitted 2009-01-20; First posted 2009-01-21 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Acute Lung Injury
Keywords: Single Nucleotide Polymorphism; cardiopulmonary bypass; cardiac surgery
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 3ml blood before surgery, after surgery and 24h after surgery respectively
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ALI: patients with acute lung injury at 24h after cardiac surgery
- Control: patients without acute lung injury 24h after cardiac surgery

SUMMARY:
Acute lung injury is a common complication of cardiac surgery with cardiopulmonary bypass, and it is significantly related to prolonged postoperative recovery, hospital stays and medical cost. Currently available predictors of acute lung injury after cardiac surgery are still limited within clinical data. Several genetic polymorphism of inflammatory mediators have been reported to be associated with severity of sepsis and ARDS, but the association of these inflammatory polymorphism and acute lung injury after cardiac surgery has never been reported. This study is performed to investigate the association of genetic polymorphisms including TNF -308A/G, IL-10 -1082A/G and IL-6 -572C/G and postoperative lung injury.

ELIGIBILITY:
Inclusion Criteria:

* Chinese Han unrelated population
* adult patients
* undergoing elective cardiac surgery with CPB

Exclusion Criteria:

* malignant tumor
* autoimmune disease, immunodeficiency or immunosuppressive therapy
* chronic renal disease (glomerular filtration rate < 60ml/(min•1.73m2)) or liver dysfunction (Child Pugh classification>A)
* COPD, tuberculosis or other chronic pulmonary diseases
* anemia with hemoglobin lower than 90mmHg
* bleeding disorders
* postoperative pericardial tamponade requiring re-operation
* postoperative low cardiac output syndrome or acute pulmonary edema after left cardiac failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unrelated Chinese Han patients undergoing elective cardiac surgery with CPB
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2008-05; Primary Completion 2008-11 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Acute lung injury after cardiac surgery with cardiopulmonary bypass | 24h after surgery

SECONDARY OUTCOMES:
circulating level of CRP, TNF-alpha, IL-10, IL-6; APACHE Ⅱ score; postoperative kidney injury, duration of ventilation, ICU stay and hospitalization; death in 28 days | 24h and 1 month after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China

REFERENCES:
- [Result] Wang JF, Bian JJ, Wan XJ, Zhu KM, Sun ZZ, Lu AD. Association between inflammatory genetic polymorphism and acute lung injury after cardiac surgery with cardiopulmonary bypass. Med Sci Monit. 2010 May;16(5):CR260-5. PMID 20424554